CLINICAL TRIAL: NCT03111849
Title: Prevalence of Sarcopenia in Chronic Obstructive Patients Hospitalized in Pneumology at the CHU of Clermont-Ferrand
Brief Title: Sarcopenia in COPD Patients: a French Study
Acronym: SARCOBS
Status: Completed | Type: Observational
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Other Study IDs: CHU-315; IRB00008526 (Other: IRB00008526)
Record Dates: First submitted 2017-04-07; First posted 2017-04-13 (Actual); Last update posted 2018-07-26 (Actual); Status verified 2018-07

CONDITIONS: COPD
Keywords: COPD; Sarcopenia; Prevalence; Mortality; Malnutrition; Nutritional assessment; Body composition; Pulmonary cachexia
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Sarcopenia; Malnutrition

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- hospitalized chronic obstructive patients
  Interventions: Other: sarcopenia

INTERVENTIONS:
Other: sarcopenia — Prevalence of sarcopenia in hospitalized chronic obstructive patients

SUMMARY:
The prevalence of sarcopenia is high in many organ pathologies such as COPD, but remains little studied in acute respiratory failure. Sarcopenia is a health problem representative of frailty, loss of autonomy and decreased muscle strength. The frequency and evolution of sarcopenia is unknown in patients having chronic bronchic obstruction with exacerbation.

DETAILED DESCRIPTION:
* Investigator consecutively included patients with known persistent airflow obstruction, hospitalized in Pneumology Department at the CHU Gabriel Montpied in Clermont-Ferrand.
* Investigator offered to participate to an observational study involving nutritional evaluation (recommended by national and international authorities) complementary to their usual respiratory care, and a 6 months' follow-up consultation: examination and surveys, mid-arm muscle circumference, body composition, spirometry.
* This enables to assess sarcopenia as a low mid-arm muscle area, by measuring the mid-arm muscle circumference of the dominant side and the triceps skinfold thickness.
* The primary endpoint is to determine the prevalence of sarcopenia, via the brachial muscular circumference, of chronic obstructive patients hospitalized in Pneumology department.
* The data entry (clinical, biological and radiological) is carried out on site, during the initial consultation and follow-up, directly on the computerized patient file. These data will then be retrieved and entered in an Excel spreadsheet, anonymously (anonymous identification number, gender and age).
* Management of censored data (lost to follow-up, cessation or withdrawal of study): each patient has a "computerized patient record" with phone numbers, checked during the first consultation and updated if necessary. The patient is called back one month before the follow-up consultation to confirm the appointment. If it is impossible to come, the patient will be offered another appointment, within one month of his initial appointment.
* Lost participants will not be excluded from statistical analyses.
* The expected number of subjects is 50.
* Oral and written consent is asked at the beginning of the consultation proposing participation in the study and follow-up at 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* A history of persistent airflow obstruction (a post-bronchodilator FEV1/FVC < 0.7 of the predicted value after 400 ug of inhaled salbutamol) compatible with respiratory function tests (according to the GOLD definition)
* Informed consent to examination of nutritional status

Exclusion Criteria:

* Bronchopulmonary cancer being treated
* Disabling rheumatic disease
* Recent stroke or surgery (< 3 months)
* Missing data on essential variables (BMI, mid-arm muscle circumference)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: chronic obstructive patients
Sampling Method: Non-Probability Sample
Enrollment: 54 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2017-10-31 (Actual); Study Completion 2017-11-30 (Actual)

PRIMARY OUTCOMES:
Prevalence of sarcopenia in hospitalized chronic obstructive patients | at day 1

SECONDARY OUTCOMES:
Evolution of sarcopenia after hospitalization | at day 1
Determination of the factors influencing this evolution | at day 1
Determination of phenotypes from anthropometric, functional and nutritional biological parameters | at day 1

CONTACTS AND LOCATIONS:
Overall Officials: Annick GREIL, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU Clermont-Ferrand, Clermont-Ferrand, France